Effects of exercise training in patients with atrial fibrillation and Sleep

apnea: A pilot study

PI: Hady Atef

Lecturer of physical therapy for cardiovascular/respiratory disorders and geriatrics

Contacts: <u>hady612@hotmail.com</u>, +2 (111-96-991-0)

## **Informed consent form**

I am freely voluntarily consenting to participate in this research study under the supervision of researcher: Hady Atef. A description of the study dates (starting 01/2019) and procedures has been explained to me and I understand that I may withdraw my consent and discontinue participation in this research study at any time without prejudice to me.

Participant name:

Signature:

Date: /1/2019